CLINICAL TRIAL: NCT04261374
Title: The Analysis of the Sublingual Microvascular Terminal Circuit Improves the Diagnostic and Therapeutic Algorithms in Dehydrated Older Patients- a Prospective Observational Study
Brief Title: Microcirculation in Dehydrated Older Patients
Acronym: MicroCirc
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: 16-003
Record Dates: First submitted 2020-01-29; First posted 2020-02-07 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Dehydration
Keywords: Microcirculation; dehydration; risk stratification
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measurement of sublingual microcirculation
  Interventions: Diagnostic Test: Measurement of sublingual microcirculation

INTERVENTIONS:
Diagnostic Test: Measurement of sublingual microcirculation — Measurement of sublingual microcirculation

SUMMARY:
This proof-of-concept study examines whether 1) sublingual measurement in dehydrated old patients is feasible, 2) frailty and incompliance in old, awake patients affects video-quality, 3) dehydration impacts microcirculation This prospective observational study includes clinically dehydrated patients aged ≥ 65 years, who have spontaneous circulation and access to the sublingual mucosa, immediately after admission. Dehydration will be assessed clinically. A sidestream dark field camera (SDF) will be used for measurement. Video-quality will be evaluated with MIQS (microcirculation image quality score). Both AVA 4.3C- and AVA POEM-software analyzed the videos. Seventeen patients ≥ 65 years not showing dehydration served as control.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* diagnosed with dehydration according to the clinical impression of the treating physician
* informed consent
* the sublingual mucosa had to be accessible.

Exclusion Criteria:

* <65 years
* Lacking informed consent
* time-critical disease
* previous resuscitation
* inaccessibility of sublingual area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who clinically dehydrated
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Percentage of Perfusion Vessels [%] | at Baseline and after 24 hours
  Measurement of sublingual microcirculation by using MicroScan® microscope. AVA 4.3C calculates automatically important microcirculatory values (Percentage of Perfusion Vessels; DeBackerDensity; Perfused DeBackerDensity; Perfused Vessel Density) according to the Second Consensus Conference

SECONDARY OUTCOMES:
Microcirculatory quality score (MIQS) | at Baseline
  MIQS by Massey et al. is an established method to validate recorded SDF-videos for their suitability for further analysis. MIQS assigns a score of optimal (0 points), suboptimal but acceptable (1 point), or unacceptable (10 points) to the categories illumination, duration, focus, content, stability, and pressure. The scoring will be done for every recorded video during the offline analysis
Clinical Frailty Scale | at Baseline
  The Clinical Frailty Scale (CFS) is a simple model visually describing patients physical conditions with nine classes from very fit (class 1) to terminally ill (class 9)
Barthel scoring | at Baseline
  Nursing status will be estimated by the Barthel-Index ranging from 100 points ("normal and autonomous") to 0 points ("completely depending from nursing").
Mini-Mental-Test scoring | at Baseline
  The standardized Mini-Mental-Test 30 is a screening tool for cognitive impairment. The test will be performed directly before SDF-measurement. The best possible result is 30 points, the worst 0 points. Test results up to 24 points can be considered normal
Rate of mortality | 30 days after discharge
  30 days mortality will be assessed using the medical records of the hospital or direct contact to the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided